CLINICAL TRIAL: NCT04886544
Title: A Multicenter, Randomized, Evaluator-Blinded, No-Treatment Control Design Clinical Study to Evaluate the Effectiveness and Safety of YVOIRE Y-Solution 720 Injected for Jawline Contouring
Brief Title: Clinical Study to Evaluate the Effectiveness and Safety of YVOIRE Y-Solution 720 Injected for Jawline Contouring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LG Chem (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LG-HACL025
Record Dates: First submitted 2021-05-10; First posted 2021-05-14 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Jaw Volume Deficit

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Experimental): Hyaluronic acid dermal filler at Week 0
  Interventions: Device: YVOIRE Y-Solution 720
- Control group (No Intervention): Remain untreated until Week 26

INTERVENTIONS:
Device: YVOIRE Y-Solution 720 — Hyaluronic acid dermal filler
  Arms: Test group

SUMMARY:
A Multicenter, Evaluator-Blinded, No-Treatment Control Design Clinical Study to Evaluate the Effectiveness and Safety of YVOIRE Y-Solution 720 Injected for Jawline Contouring

DETAILED DESCRIPTION:
This is a Multicenter, Randomized, Evaluator-Blinded, No-Treatment Control Design Clinical Study to Evaluate the Effectiveness and Safety of YVOIRE Y-Solution 720 Injected for Jawline Contouring.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults 18 - 75 years of age (inclusive)
* 2 (moderate) or 3 (severe) on Jawline Contour Rating Scale (JCRS)
* want a filler injection procedure for the replacement of volume loss in the jawlines

Exclusion Criteria:

* have an active or infective skin disease
* have lower-face volume deficit due to congenital defect, trauma, abnormalities in adipose tissue related to immune-mediated diseases
* have a tattoo or excessive facial hair in the evaluation area
* have received permanent facial implants
* have undergone semi-permanent filler within 24 months
* have undergone temporary dermal filler treatment in the lower face (below the orbital rim) within 12 months
* have streptococcal disease
* have a medical history of hypertrophic cicatrix, hyperpigmentation or keloid
* have a history of anaphylaxis, multiple severe allergies, or allergy to lidocaine (or any amide-based anesthetic), or hyaluronic acid products
* have history of bleeding disorder
* have severe cardiovascular, hepatic or renal diseases considered as per Investigator's discretion
* have known malignant tumors or cancerous or precancerous lesion
* positive pregnancy test indicating pregnancy
* active COVID-19 infection and suspected COVID-19 infection within the past 14 days

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2021-06-25 (Actual); Primary Completion 2022-05-11 (Actual); Study Completion 2023-01-09 (Actual)

PRIMARY OUTCOMES:
The primary effectiveness endpoint is the Jawline Contour Rating Scale (JCRS) responder rate at 26 weeks after the last injection | 26 weeks from baseline
  The primary effectiveness endpoint is the Jawline Contour Rating Scale (JCRS) responder rate at 26 weeks after the last injection for the test group and at Week 26 for the control group, i.e., the proportion of subjects with ≥1 grade improvement on the JCRS score (both jawlines) rated by independent blinded Evaluators at the site (Evaluating Investigator) at Visit 5, compared to that at Baseline (Visit 1).

CONTACTS AND LOCATIONS:
Overall Officials: Principal Investigator, Principal Investigator — LG Chem Investigational site 01
Locations (3):
- Austria (2):
  - LG Chem investigational site 01, Vienna
  - LG Chem investigational site 02, Vienna
- LG Chem investigational site 03, Krakow, Poland